CLINICAL TRIAL: NCT03070821
Title: Neurofeedback and Follow-up With Real-time fMRI to Investigate Cognitive Function in Patients of Mild Cognitive Impairment (MCI) or Alzheimer's Disease (AD)
Brief Title: Therapy of Alzheimer's Disease With Neurofeedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Aachen (Other)
Collaborators: Alzheimer Forschung Initiative e.V. (Unknown)
Responsible Party: Principal Investigator, Kathrin Reetz, Head of Memory Clinic and/or Principal Investigator, University Hospital, Aachen
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFI 13812
Record Dates: First submitted 2017-02-23; First posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-02

CONDITIONS: Alzheimer Dementia (AD); Elderly
Keywords: neurofeedback; real-time functional MRI; parahippocampus
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The design is a pre-test/post-test study with an intervention of three parallel groups. The groups are a healthy elderly experimental group, a patient group and a healthy elderly sham-feedback group.
Who Masked: Participant
Masking Description: Healthy subjects in the sham feedback condition were not aware of their group membership, but were debriefed at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy elderly experimental group (Experimental): Feedback of the parahippocampal gyrus using rtfMRI neurofeedback training (using 3T MRI).
  Interventions: Other: rtfMRI neurofeedback training; Device: 3T MRI
- Patient group (Experimental): Feedback of the parahippocampal gyrus using rtfMRI neurofeedback training (using 3T MRI).
  Interventions: Other: rtfMRI neurofeedback training; Device: 3T MRI
- Healthy elderly sham-feedback group (Sham Comparator): Feedback of the postcentral gyrus using rtfMRI neurofeedback training (using 3T MRI).
  Interventions: Other: rtfMRI neurofeedback training; Device: 3T MRI

INTERVENTIONS:
Other: rtfMRI neurofeedback training — Information about the state of brain activation was given to subjects. That information was visualised as a thermometer bar. Subjects tried to modulate that activation while performing a mental imagery task.
Device: 3T MRI — A 3T Siemens MRI scanner was used to implement rtfMRI neurofeedback training.

SUMMARY:
The project aims to investigate in patients of Alzheimer's disease in a prodromal state (early state of the disease) compared to healthy subjects whether neurofeedback training with functional MRI (fMRI) can improve cognitive ability. It is of interest if voluntary modulation of brain activation with real-time (rt) fMRI as a novel method affects cognitive ability, as well as functional and structural measures of the brain.

Over the course of the study subjects will learn a real-world footpath. During neurofeedback training subjects are then asked to recall this footpath while simultaneously trying to modulate their own brain activation based on feedback. Feedback is given about the parahippocampal gyrus - a region of the brain associated with episodic and visuo-spatial memory, which is known to be affected early by Alzheimer's disease pathology.

Before and after the training cognitive ability is assessed using neuropsychological tests mainly measuring numerous domains of memory.

The investigators hypothesise that the training leads to an improvement of the trained cognitive domain, but also induces changes in brain structure and function.

ELIGIBILITY:
Inclusion Criteria:

* Native speakers of German
* Naive to neurofeedback experiments
* Ability to provide written informed consent

Exclusion Criteria:

* Metallic implants (MR-safety)
* Neurological/psychiatric disease (except Alzheimer's disease in the patient group)
* Use of psychoactive medication (expect medication for Alzheimer's disease)
* Familiarity with the study site

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01-30 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Visual and Verbal Memory Test (VVM) | 2.5 weeks
  Neuropsychological assessment including visuo-spatial memory

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 2.5 weeks
  Neuropsychological instrument for a general cognitive screening
Wechsler Memory Scale Revised (WMS-R) | 2.5 weeks
  Subtests from the WMS-R were used to assess several domains of memory
Trail Making Test (TMT) | 2.5 weeks
  TMT-A and -B were used to assess cognitive processing speed and task switching capabilities.
Visual Patterns Test (VPT) | 2.5 weeks
  The VPT was used to assess visual working memory capabilities.
Parahippocampal activation | 2.5 weeks
  Activation of the parahippocampal gyrus during neurofeedback training as measured with fMRI
Memory-related functional connectivity using Granger Causality Analysis (GCA) | 2.5 weeks
  Change of functional connectivity mainly between memory-associated brain regions over the course of neurofeedback training characterised by GCA
Change of brain structure | 2.5 weeks
  Assessment of grey matter volume in the entire brain
Change of brain function | 2.5 weeks
  Assessment of activation in the entire brain

CONTACTS AND LOCATIONS:
Overall Officials: Kathrin Reetz, Prof. Dr., Principal Investigator — University Hospital, Aachen

IPD SHARING:
Plan to Share IPD: No